CLINICAL TRIAL: NCT03837405
Title: Optimizing Lifestyle Interventions With Mindfulness-based Strategies in Type 2 Diabetes
Brief Title: (R33 Phase) Delish Study: Diabetes Education to Lower Insulin, Sugars, and Hunger
Acronym: Delish R33
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4R33AT009333 (NIH); 4R33AT009333 (NIH)
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blood tests at LabCorp and 24-hour dietary recall interviews are done by research assistants blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Education (Active Comparator): All participants will receive instruction in the Carbohydrate-Restricted (CR) diet and basic behavioral strategies in weekly, in-person, group sessions for 3 months. The study diet has approximately 10% of kcal coming from carbohydrate, typically 50 grams/day or fewer, not including fiber. Participants will be encouraged to eat a normal amount of protein, typically about 80-100 grams/day (about 20-25% of calories), and the rest of their calories from fat.
  Interventions: Behavioral: Carbohydrate-restricted diet
- Diet Education + Mindfulness (Experimental): In addition to the diet components described above, participants randomized to the Education + Mindfulness (Ed+MBI) group will receive MBI components using the Eat Right Now (ERN) platform. This will consist of two integrated components: 1) use of the ERN app at home, during the week, to learn and practice mindfulness skills for food-cravings and eating, and 2) in-person group-based discussions of how the mindful eating practices are going, trouble-shooting obstacles/pain points, and doing group exercises and reflecting on them.
  Interventions: Behavioral: Carbohydrate-restricted diet; Behavioral: Mindfuless

INTERVENTIONS:
Behavioral: Carbohydrate-restricted diet — Education for carbohydrate-restricted diet
Behavioral: Mindfuless — Mindful eating app use plus group sessions to learn mindfulness
  Arms: Diet Education + Mindfulness

SUMMARY:
The investigators plan an R33 phase trial in which 120 persons with type 2 diabetes (T2DM) will be randomized (using a 1:1 ratio) to education alone (Ed) on following a carbohydrate restricted diet for T2DM, or this same education content with added mindful eating/Mindfulness-Based Intervention components (Ed+MBI).

DETAILED DESCRIPTION:
The investigators will randomize 120 persons with T2DM in a 1:1 ratio to a nutrition education alone arm (Ed n=60) vs. a nutrition education with mindfulness-based intervention components (Ed+MBI n=60) arm and follow them for 12 months. The interventions will be provided in a weekly group setting, with about 10 to 12 persons per group. Some educational intervention components will be delivered using a smartphone app. After the 12-week initial intervention, the investigators will re-randomize participants using an adaptive intervention design to receive low, medium, or high intensity maintenance training, depending on level of adherence achieved during the initial intervention period. Follow-up assessments will be performed at 3, 6, 9, and 12 months. The investigators will address the following specific aims:

1. Test the hypothesis that the Ed+MBI arm will have better dietary adherence than the Ed arm.
2. Test whether our proposed behavioral mechanisms (e.g. decreased eating in response to cravings or difficult emotions) predict dietary adherence.
3. Compare randomized arms in the adaptive maintenance intervention design to optimize maintenance phase dosing in future trials.
4. Obtain preliminary assessment of intervention effects on clinical outcomes

This is the second phase of a two-phase study. Pilot testing has been completed in the first phase (R61). The second phase (R33) will include employing an adaptive intervention design in the post-treatment phase to test optimization of the maintenance intervention (i.e. assigning maintenance intensity/dose based on how a participant is doing). The investigators will use fingerstick blood ketone measures, which provide an objective measure of whether the target levels of carbohydrate restriction have been attained, as our primary adherence outcome measure. This will be supplemented by 24-hour diet recall measures of carbohydrate consumption. Important secondary outcome measures will include clinical measures such as glycosylated hemoglobin and behavioral measures such as frequency of eating in response to food cravings.

ELIGIBILITY:
Inclusion Criteria:

1. History of T2DM mellitus.
2. HbA1c ≥ 6.5% and < 12.0% at screening.
3. Experience food-related cravings most days of the week and eat in response to these cravings regularly.
4. Aged 18 years old and older.
5. Able to engage in light physical activity.
6. Willing and able to participate in the interventions including appropriate participation in the group setting.
7. Have smartphone and are willing to use it on a regular basis for data collection.
8. Ability to speak English.

Exclusion Criteria:

1. Unable to provide informed consent.
2. A substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate in the intervention, that may need immediate changes in medical management that will affect study outcome measures, or that may require important adaptations in the study diet.
3. Pregnant or planning to get pregnant in the next 12 months, breastfeeding or less than 6 months post-partum.
4. Current use of weight loss medications, such as Alli or amphetamine-based drugs that may affect weight.
5. Planned or history of weight-loss (bariatric) surgery, or other intestinal surgeries that cause malabsorption. These are likely to change study outcome measures, making it difficult to distinguish the effects of the intervention program, or require extensive tailoring of the diet intervention.
6. Currently enrolled in a weight loss program, such as Weight Watchers or a self-help group such as Overeaters Anonymous, or have unalterable plans to enroll in one of these programs in the next year; using a ketogenic low carbohydrate diet in the past 6 months with advice from a health care professional; or use of a mindful eating program with guidance from a professional in the past 6 months or have ever used the study mindful-eating app.
7. Vegan or vegetarian.
8. Unwilling to do regular blood testing at home for glucose or ketone monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
diet adherence between intervention arms as measured by ketones | measures from ketone measure initiation (week 5) to 12 months
  proportion of ketone measures dichotomized as > or = 0.3 mmol/L versus < 0.3
diet adherence between intervention arms as measured by 24- hour diet recall--dichotomous | from 3 to 12 months
  proportion of participants consuming < 50 grams/day of non-fiber carbohydrate (from 24-hour diet recall)

SECONDARY OUTCOMES:
executive functioning /decreased impulsivity-Delayed Discounting | change from baseline to 12 months
  change in Delayed Discounting task score
emotion-related eating | change from baseline to 12 months
  change in emotion-related eating as measured by the Coping subscale of the Palatable Eating Motives Scale (PEMS).
Glycemic control--a1c | change from baseline to 12 months
  hemoglobin a1c
frequency of eating in response to cravings | change from baseline to 12 months
  frequency of eating in response to cravings using ecological momentary assessment (EMA)
diet adherence between intervention arms as measured by 24- hour diet recall--total carbs, continuous | from 3 to 12 months
  mean grams of non-fiber carbohydrate consumed per day (from 24-hour diet recall)
executive functioning /decreased impulsivity--Relative Reinforcing Value of Food (RRVF) | change from baseline to 12 months
  change in RRVF score
Salzburg Stress Eating Scale | change from baseline to 12 months
  change in stress-related eating as measured by Salzburg Stress Eating Scale
dietary resilience (resumption of dietary adherence) after dietary non-adherence occurs | 12 months
  time from a ketone measure of < 0.3 mmol/L to higher levels of >/= 0.3 mmol/L
Weight change | change from baseline to 12 months
  pounds

OTHER OUTCOMES:
stress-related eating | change from baseline to 12 months
  change in stress-related eating as measured by two questions about stress-related eating from the MIDUS study and one additional stress-related eating question
Perceived Stress | change from baseline to 12 months
  change in Perceived Stress Scale total score
Insulin resistance | change from baseline to 12 months
  Homeostatic model assessment (HOMA) index of insulin resistance (computed from insulin and fasting glucose measures)
Glycemic control--fasting glucose | change from baseline to 12 months
  fasting blood glucose
Mindfulness | change from baseline to 12 months
  Five-factor mindfulness scale

CONTACTS AND LOCATIONS:
Overall Officials: Rick Hecht, MD, Principal Investigator — University of California, San Francisco; Elissa Epel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03837405/ICF_000.pdf